CLINICAL TRIAL: NCT06644066
Title: Application of Partial Pressure of Oxygen Control Method in Fast Identification of Intersegmental Plane in Anatomical Sublobar Resection: a Prospective, Randomized Controlled Study
Brief Title: Partial Pressure of Oxygen Control Method in Identification of Intersegmental Plane
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K202406-24
Record Dates: First submitted 2024-07-01; First posted 2024-10-16 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Lung Cancer
Keywords: Sublobar resection; Intersegmental plane; Non small cell lung cancer(NSCLC); Partial pressure of Oxygen Control method; Video-assisted thoracoscopic(VATS)
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partial pressure of Oxygen Control method (Experimental): After the targeted structures were successfully dissected, the anesthesiologist manually controls pure oxygen one-lung ventilation on the surgical side until the lung is fully expand. The ventilator is disconnected, the airway is opened, and the operator uses a gauze ball to pressure the preserve lung tissue. At a SpO2 of 95%, the healthy side undergoes one-lung ventilation.
  Interventions: Procedure: Partial pressure of Oxygen Control method
- Modified inflation-deflation method (No Intervention): After the targeted structures were successfully dissected, and then the collapsed lung was re-expanded completely with controlled airway pressure under 20 cmH2O, with the bronchus of the operation side open to atmosphere while continuing ventilation of the contralateral lung.

INTERVENTIONS:
Procedure: Partial pressure of Oxygen Control method — During the process of inflation-deflation, by maintaining a lower PaO2, the identifying the intersegmental plane is accelerated
  Arms: Partial pressure of Oxygen Control method

SUMMARY:
In recent years, an increasing number of pulmonary nodules have been detected through CT screening. The traditional surgical method for lung cancer is lobectomy combined with lymph node dissection. However, recent studies have demonstrated that sublobar resection for early non-small cell lung cancer (NSCLC) is an effective alternative with the additional benefit of preserving more pulmonary function. However, it also faces many problems, the most prominent of which is the rapid and accurate identification of the intersegmental plane (ISP) during surgery. The modified inflation-deflation method for identifying the ISP is the most commonly used method in anatomical sublobar resection. Nevertheless, the lengthy waiting periods and the lack of clear delineation represent significant challenges in clinical practice. The Partial pressure of Oxygen Control method facilitates the efficient determination of the ISP by reducing the oxygen inhalation concentration and ventilator ventilation time during surgery. This results in a reduced PaO2 in arterial blood, thereby accelerating the rapid appearance of the ISP. Thus, the investigators conducted a prospective, randomized, controlled trial to ascertain whether the oxygen partial pressure control method affects the occurrence time of the ISP and PaO2 during one-lung ventilation, in comparison to the modified inflation-deflation method. Furthermore, the objective was to confirm the safety and efficacy of Partial pressure of Oxygen Control method.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 75;
2. Gender unlimited;
3. Eastern Cooperative Oncology Group（ECOG） Performance status（PS） score 0-1 points;
4. Thin slice CT indicates that the maximum tumor diameter is ≤ 2.0cm and 0 ≤ CTR<1.0; （Consolidation Tumor Ratio，CTR）
5. Those who voluntarily sign the informed consent form for research can comply with the requirements of the research visit plan and other protocols.

Exclusion Criteria:

1. Individuals with a history of lung surgery in the past;
2. Patients with interstitial pneumonia, pulmonary alveoli, pulmonary fibrosis, or severe emphysema;
3. Those who undergo chest surgery due to various reasons or change the surgical plan during the operation;
4. The subjects do not understand, cooperate or refuse to sign the informed consent form regarding the research protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Time of Intersegmental plane（TISP） | Throughout the entire surgical period，an average of 10 minutes
  The start time was defined as the end of the surgical side lung having completely re-expanded. The end point was identified as the point at which the preserved lung was fully deflated, and a boundary had formed between the targeted lung tissue and the reserved lung.
The lung collapse score | Throughout the entire surgical period
  The lung collapse score was referenced and improved by the Bussiers method using descriptive and visual features that included the context of lung collapse, space in the thermal cavity, atelectasis, color of the lung (healthy lungs are a pink gray/simple color), and where the collapse was considered satisfactory.Lung collapse was defined on a 4-point scale, where 1 point int=no lung collapse, 2 point=less partial lung collapse, 3 point=major partial lung collapse, 4 point=total lung collapse Each video clip was assessed by 2 evaluators。 Independently evaluate the level, and resolve differences through consensus through negotiation.

SECONDARY OUTCOMES:
Surgical time | Throughout the entire surgical period，An average of 120 minutes
  The total time from the start of skin incision to the completion of chest closure
Blood gas analysis | Throughout the entire surgical period，Baseline, Up to 120 minutes
  Blood gas analysis measuring before entry, after one lung ventilation (SpO2 maintained at 95%), after pure oxygen lung stimulation, and at 3 and 6 minutes after pure oxygen lung expand.
Intraoperative bleeding volume | Throughout the entire surgical period
  Intraoperative bleeding volume: Use a suction device and a graduated collection device to collect intraoperative bleeding volume in milliliters, accurate to ten digits. (An average of 50ml)
Postoperative drainage volume | Intraoperative
  Postoperative drainage volume: The total drainage volume in the drainage bottle during the retention of the thoracic catheter after surgery, in milliliters. (An average of 200ml)
Postoperative complication incidence | Throughout the perioperative period，Baseline, Up to 3 months
  Postoperative complication incidence: Record the name of the complication and classify it according to the Clavien Indo classification system
Postoperative hospitalization days | From surgery to discharge ，An average of 5 days
  The number of days between the surgical date and the discharge date;
Total hospitalization cost | Up to 3 months
  Total hospitalization cost: The total cost of patients from admission to discharge, settled in ChiNaYuan（CNY） (before medical insurance settlement).

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of the Air Force Medical University of PLA, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Xing M, Tong L, Duan H, Aliev D, Dong X, Zhang Y, Liu H, Yan X. Partial pressure of oxygen control versus modified inflation-deflation method in identifying intersegmental plane during anatomical sublobectomy: a prospective, randomized, controlled trial. J Thorac Dis. 2025 Feb 28;17(2):1042-1053. doi: 10.21037/jtd-2025-45. Epub 2025 Feb 27. PMID 40083504